CLINICAL TRIAL: NCT02794142
Title: Impact of the Oxidative Stress on the Skeletal Muscle Dysfunction in Hemodialysis Patient
Brief Title: Oxidative Stress on Muscle Dysfunction in Hemodialysis Patient
Acronym: POPEYE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9459-2
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Chronic Renal Failure Requiring Hemodialysis
Keywords: hemodialysis; muscle dysfunction; mitochondria; oxidative stress; inflammation; renal transplantation
MeSH Terms: conditions — Inflammation | interventions — Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HD patient (Experimental)
  Interventions: Procedure: renal transplantation
- Healthy volunteers (Other)
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: renal transplantation
  Arms: HD patient
Other: No intervention
  Arms: Healthy volunteers

SUMMARY:
In hemodialysis patient (HD) a reduction of the skeletal muscle mass and strength has previously been reported. This muscle impairment constitutes an independent prognosis factor in HD patients. Oxidative stress and inflammation have been linked to the muscle impairment. The mitochondria is a classical producer and target of reactive oxygen species (ROS), and may thus constitute a central actor of the skeletal muscle impairment in HD patients. Therefore, the aim of the present study is to investigate the role of the muscle mitochondrial density on the muscle impairment in HD patients, in comparing the muscle mitochondrial density and oxidative stress in HD patients vs. healthy matched controls.

In order to assess the effect of the oxidative stress and inflammation on the muscle impairment in HD patients, muscle function assessements will be performed after renal transplantation (which lowers the oxidative stress and inflammation levels) in the HD patient group.

No therapeutic intervention will be tested in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-80 years old
* less than 150min by week of moderate to vigorous physical activity
* Chronic renal failure (glomerular filtration rate less than 15mL by min) requiring hemodialysis
* Patient placed on the kidney transplant waiting list of MontpellierCHU
* No indication against temporary kidney transplant
* Review cardiovascular older than two years
* Patient not under guardianship or trusteeship
* Clinically stable state Absence or recent infection within 3 months prior to inclusion Absence of progressive neoplasia No recent acute decompensation of chronic disease (thrust of heart failure, respiratory decompensated cirrhosis).

Absence of recent stroke

* musculoskeletal and neurological states of the lower limbs which allow the realization of the proposed functional tests.
* Patient has given written informed consent
* Absence of congenital or genetic degenerative muscle disease

Exclusion Criteria:

* Terminal chronic renal failure without replacement therapy
* Local anesthesic hypersensibility
* Corticosteroid treatment upper than 3 month
* COPD
* Oral anticoagulants
* Previous renal transplantation
* Subject not affiliated with a social security scheme, beneficiary or not such a plan
* Major subject protected by law or unable to consent under Article L 1121-8 of the Public Health Code
* Vulnerable person under Article L.1121-6 of the Public Health Code

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Muscle mitochondrial density assessed on a quadriceps biopsy by immunochemistry | 2 years

SECONDARY OUTCOMES:
Maximum voluntary contraction of the quadriceps (in Newton.meter) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

REFERENCES:
- [Derived] Souweine JS, Gouzi F, Badia E, Pomies P, Garrigue V, Morena M, Hayot M, Mercier J, Ayoub B, Quintrec ML, Raynaud F, Cristol JP. Skeletal Muscle Phenotype in Patients Undergoing Long-Term Hemodialysis Awaiting Kidney Transplantation. Clin J Am Soc Nephrol. 2021 Nov;16(11):1676-1685. doi: 10.2215/CJN.02390221. PMID 34750160